CLINICAL TRIAL: NCT01253928
Title: Effects of Pioglitazone on Body Composition,Insulin Sensitivity and Protein Metabolism in ESRD Non Diabetic Individuals
Brief Title: Pioglitazone, Body Composition,Insulin Sensitivity and Protein Metabolism in ESRD
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire Vaudois (Other)
Responsible Party: Anne Zanchi MD, CHUV
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 224/05
Record Dates: First submitted 2010-12-03; First posted 2010-12-06 (Estimated); Last update posted 2010-12-06 (Estimated); Status verified 2007-02

CONDITIONS: ESRD
Keywords: body composition; insulin sensitivity; protein metabolism; pioglitazone
MeSH Terms: conditions — Kidney Failure, Chronic; Insulin Resistance | interventions — Pioglitazone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Pioglitazone 45mg per day (Active Comparator): Pioglitazone 45mg qd will be added to the current treatment
  Interventions: Drug: Pioglitazone
- placebo (Placebo Comparator): placebo qd will be added to current treatment
  Interventions: Drug: Pioglitazone

INTERVENTIONS:
Drug: Pioglitazone — 45mg qd for 4 months
  Other Names: Actos 45mg P05W8

SUMMARY:
Non diabetic patients on renal replacement therapy are prone to changes in body composition with an increase in visceral fat and muscle wasting all favoured by the insulin resistant state. Malnutrition is associated with a worst prognosis in these patients. Glitazones are the most powerful insulin sensitisers available in clinical practice which also have anti-inflammatory properties. Their use has been associated with significant and favourable changes in body fat distribution in type 2 diabetic subjects. Experimental studies suggest that glitazones may attenuate muscle wasting in renal failure.

The goal of this study was to examine in non diabetic ESRD patients the effects of pioglitazone on inulin sensitivity and protein metabolism as determined by the hyperinsulinemic euglycemic clamp and on changes in body composition as determined by anthropometric measurements, dual energy X-ray absorptiometry (DEXA) and CT-scan determined changes in abdominal visceral and sub-cutaneous fat.

ELIGIBILITY:
Inclusion Criteria:

Non diabetic individuals with ESRD, on hemodialysis or peritoneal dialysis for at least 3 months. Consent form signed -

Exclusion Criteria:

No infectious complication 3 months prior to entry in the study.

-

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2007-03; Primary Completion 2011-06 (Estimated)

PRIMARY OUTCOMES:
Body composition | at the end of each treatment phase (which lasts 4 months)
  Effect of pioglitazone on the body composition determined by DEXA, abdominal CT, anthropometric measurements.
Insulin sensitivity | at the end of each treatment phase (which lasts 4 months)
  Hepatic and whole body insulin sensitivity will be determined during the insulin glucose clamp.
Protein metabolism | at the end of each treatment phase (which lasts 4 months)
  Protein turnover will be determined by leucine infusion during the insulin glucose clamp

CONTACTS AND LOCATIONS:
Overall Officials: Anne Zanchi, MD, Principal Investigator — CHUV Lausanne
Locations (1):
- Nephrology Service Department of Medicine CHUV, Lausanne, Canton of Vaud, Switzerland

REFERENCES:
- [Derived] Zanchi A, Tappy L, Le KA, Bortolotti M, Theumann N, Halabi G, Gauthier T, Mathieu C, Tremblay S, Bertrand PC, Burnier M, Teta D. Pioglitazone improves fat distribution, the adipokine profile and hepatic insulin sensitivity in non-diabetic end-stage renal disease subjects on maintenance dialysis: a randomized cross-over pilot study. PLoS One. 2014 Oct 16;9(10):e109134. doi: 10.1371/journal.pone.0109134. eCollection 2014. PMID 25330088